CLINICAL TRIAL: NCT00818337
Title: Aspirin Responsiveness in Women at Risk for Cardiac Events: A Pilot Study.
Brief Title: Aspirin Responsiveness in Women at Risk for Cardiac Events
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 08-14888
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aspirin 81mg (Active Comparator): Resistant
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin 81mg and Aspirin 325mg, non-enteric coated, take one tablet by mouth daily

SUMMARY:
The objective of this pilot study is to evaluate the prevalence of biological aspirin resistance in women at risk for CHD taking low dose (81 mg) aspirin. Aspirin responsiveness will be measured with the VerifyNow device (Accumetrics; San Diego, CA). Those women identified as biologically resistant will be switched to aspirin 325 mg for 14 days and then re-tested for aspirin responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 19 years old
* Taking 81 mg aspirin daily, non-enteric coated, for at least one month for the primary prevention of cardiovascular disease.
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Known CHD
* Currently taking clopidogrel or ticlopidine
* Use of heparin, warfarin, or glycoprotein IIb/IIIa inhibitors within previous 96 hours
* Allergy or hypersensitivity to salicylates
* Use of other OTC or prescription analgesics or anti-inflammatory medication in the past two weeks
* Currently participating in another investigational drug or device study

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Cardiac Center at Creighton University, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin 81mg: Aspirin 81mg at baseline
Period: Overall Study
Arm/Group | Aspirin 81mg
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aspirin 81mg
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years]
  Non-resistant to 81 mg | 52.6 (8.3)
  Resistant to 81 mg | 56.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Aspirin Resistant
Description: Aspirin responsive unit (ARU) > 550 was considered to be aspirin resistant and correlates to less than 50% inhibition of platelet aggregation.
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Aspirin 81 mg: Aspirin 81 mg at baseline
Arm/Group | Aspirin 81 mg
Number analyzed (Participants) | 36
participants | 3

2. Secondary Outcome: Number of Aspirin Resistant Who Became Responders After Increase to Aspirin 325 mg
Description: Aspirin resistance was defined as ARU > 550
Time Frame: 2 weeks
Measure: Number; unit: participants
Groups:
- Aspirin 325 mg: Participants who were aspirin resistant who were increased to aspirin 325 mg
Arm/Group | Aspirin 325 mg
Number analyzed (Participants) | 3
participants | 3

ADVERSE EVENTS:
Arm/Group | Aspirin 81mg
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes